CLINICAL TRIAL: NCT02926690
Title: A Phase I Study of OTS167PO, a MELK Inhibitor, to Evaluate Safety, Tolerability and Pharmacokinetics in Patients With Advanced Breast Cancer and Dose-Expansion Study in Patients With Triple Negative Breast Cancer
Brief Title: Safety Study of MELK Inhibitor to Treat Patients With Advanced Breast Cancer and Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OncoTherapy Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTS1070103
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-03

CONDITIONS: Relapsed/Refractory Locally Advanced or Metastatic Breast Cancer and Triple Negative Breast Cancer
MeSH Terms: conditions — Recurrence; Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OTS167PO (Experimental)
  Interventions: Drug: OTS167PO

INTERVENTIONS:
Drug: OTS167PO — Single arm, no competitor

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of OTS167 administered via oral capsule (PO) to patients with relapsed/refractory locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation and Dose Expansion Cohorts

Patients must meet all of the following criteria to be eligible for participation in the study:

1. Female patients, ≥ 18 years of age at the time of obtaining informed consent.
2. Patients with a documented (histologically- or cytologically-proven) breast cancer that is locally advanced or metastatic.
3. Patients with a malignancy that is either relapsed/refractory to standard therapy or for which no standard therapy is available.
4. Patients with a malignancy that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
5. Patients with measurable or non-measurable disease according to the Response Evaluation Criteria In Solid Tumor (RECIST, v1.1).
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 (see APPENDIX B: Performance Status Evaluation).
7. Life expectancy of greater than or equal to 3 months.
8. Resolution of all chemotherapy-related or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (less than or equal to Grade 2).
9. Patients who are either not of childbearing potential or who agree to use a medically effective method of contraception during the study and during 3 months after the last dose of study drug. (See Appendix H: Forms of contraception).
10. Patients with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Dose expansion Cohort - TNBC

1. Patients with conditions as follows:

   * ER <10%, PR <10% by IHC assay; And
   * HER2 negative based on ASCO CAP guideline
2. Patients with measurable disease according to the response evaluation criteria in TNBC (RECIST, v1.1)
3. Patients with measurable disease that can be easily accessed for biopsy.
4. Relapsed (recurrence or disease progression after achieving a documented clinical response to first- or second-line treatment) or refractory (disease progression while receiving first line or second line treatment). In the case of TNBC, prior initial therapy with at least one known active regimen for TNBC including, but not limited to, any combination of anthracyclines, taxanes, platinum agents, Ixabepilone, and/or cyclophosphamide is required.

Exclusion Criteria:

Dose Escalation and Dose Expansion Cohorts Patients meeting any of the following criteria are ineligible for participation in the study.

1. Women who are pregnant or lactating. Women of child-bearing potential (WOCBP) not using adequate birth control see Appendix H: Forms of contraception.
2. Patients with known central nervous system (CNS) or leptomeningeal metastases not controlled by prior surgery, radiotherapy or requiring corticosteroids to control symptoms, or patients with symptoms suggesting CNS involvement for which treatment is required.
3. Patients with primary brain tumors.
4. Patients with any hematologic malignancy. This includes leukemia (any form), lymphoma, and multiple myeloma.
5. Patients with any of the following hematologic abnormalities at baseline. (Patients may have received a red blood cell product transfusion prior to study, if clinically warranted.):

   * Absolute neutrophil count (ANC) < 1,500 per mm3
   * Platelet count < 100,000 per mm3
   * Hemoglobin < 8.0 gm/dL
6. Patients with any of the following serum chemistry abnormalities at baseline:

   * Total bilirubin ≥ 1.5 × the ULN for the institution value
   * AST or ALT ≥ 3 × the ULN for the institution value (≥ 5 × if due to hepatic involvement by tumor)
   * Creatinine ≥ 1.5 × ULN for the institution value (or a calculated creatinine clearance < 60 mL/min/1.73 m2* )
7. Patients with a significant active cardiovascular disease or condition, including:

   * Congestive heart failure (CHF)requiring therapy
   * Need for antiarrhythmic medical therapy for a ventricular arrhythmia
   * Severe conduction disturbance
   * Unstable angina pectoris requiring therapy
   * QTc interval > 450 msec (males) or > 470 msec (females)
   * QTc interval ≤ 300 msec
   * History of congenital long QT syndrome or congenital short QT syndrome
   * LVEF < 50% as measured by echocardiography or MUGA scan
   * Uncontrolled hypertension (per the Investigator's discretion)
   * Class III or IV cardiovascular disease according to the New York Heart Association's (NYHA) Functional Criteria (see APPENDIX C: New York Heart Association's Functional Criteria).
   * Myocardial infarction (MI) within 6 months prior to first study drug administration
8. Patients with a known or suspected hypersensitivity to any of the components of OTS167.
9. Patients with a known history of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
10. Patients with any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 1 week prior to first study drug administration.
11. Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to first study drug administration.
12. Patients with any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug.
13. Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies.
14. Patients with the inability or with foreseeable incapacity, in the opinion of the Investigator, to comply with the protocol requirements.
15. Any anti-neoplastic agent or monoclonal antibody therapy for the primary malignancy (standard or experimental) within 2 weeks prior to first study drug administration.
16. Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment. If acute symptoms of radiation have fully resolved, the extent and timing of radiotherapy for eligibility can be discussed between Investigator and Sponsor.
17. Patients requiring surgery for the primary or metastatic primary malignancy.
18. Herbal preparations or related over the counter (OTC) preparations/supplements containing herbal ingredients within 1 week prior to first study drug administration and during study.
19. Systemic hormonal therapy which is not related to breast cancer treatment (standard or experimental) within 1 week prior to first study drug administration and during study. The following therapies are allowed:

    * Hormonal therapy (e.g., Megace) for appetite stimulation
    * Nasal, ophthalmic, inhaled, and topical glucocorticoid preparations
    * Oral replacement glucocorticoid therapy for adrenal insufficiency
    * Low-dose maintenance steroid therapy for other conditions (excluding steroid tapers for brain edema/metastases/radiation)
    * Hormonal contraceptive therapy (for WOCBP must be combined with non-hormonal contraceptive equivalent to a double-barrier method)
20. Any other investigational treatments during study. This includes participation in any medical device or therapeutic intervention clinical trials.

    Dose expansion Cohort - TNBC
21. Patients with only lesions that cannot be accessed for biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
MTD | During Cycle1 after the first administration

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Norwalk Hospital, Norwalk, Connecticut
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Kapi'olani Medical Center for Women & Children, Honolulu, Hawaii
  - Dartmouth Cancer Center/Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Medicine | NewYork-Presbyterian, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No